CLINICAL TRIAL: NCT05074589
Title: A Randomized, Double-blind, Single-dummy, Parallel-controlled, Multicentre, Phase III Clinical Study of Irinotecan Hydrochloride Liposome in Combination With 5-FU/LV as Second-line Treatment for Locally Advanced or Metastatic Pancreatic Cancer After Treatment Failure With Gemcitabine-based Therapy
Brief Title: Irinotecan Liposome in Combination With 5-FU/LV Versus 5-FU/LV in Second-line Therapy for Gemcitabine-Refractory Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-IRI-APC
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Second-line Treatment for Locally Advanced or Metastatic Pancreatic Cancer After Treatment Failure With Gemcitabine-based Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, single-dummy, parallel-controlled, multicentre study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Irinotecan liposome plus 5-fluorouracil, Leucovorin
  Interventions: Drug: Irinotecan liposome、5-Fluorouracil、Leucovorin
- Treatment group B (Active Comparator): Placebo plus 5-fluorouracil, Leucovorin
  Interventions: Drug: Placebo、5-Fluorouracil、Leucovorin

INTERVENTIONS:
Drug: Irinotecan liposome、5-Fluorouracil、Leucovorin — Irinotecan liposome、5-Fluorouracil、Leucovorin
  Arms: Treatment group A
Drug: Placebo、5-Fluorouracil、Leucovorin — Placebo、5-Fluorouracil、Leucovorin
  Arms: Treatment group B

SUMMARY:
To evaluate efficacy and safety of irinotecan hydrochloride liposome in combination with 5-FU/LV as second-line treatment for locally advanced or metastatic pancreatic cancer after treatment failure with gemcitabine-based therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed pancreatic cancer;
2. Unresectable locally advanced or metastatic disease ;
3. Documented disease progression after first-line treatment gemcitabine based therapy
4. ECOG: 0-1;
5. Adequate organ and bone marrow function;
6. sign an informed consent.

Exclusion Criteria:

1. Active CNS metastasis;
2. Uncontrolled tumor-related pain;
3. Clinically significant GI disorders;
4. Significant cardiovascular disease;
5. Active infection or uncontrolled fever;
6. Pregnant or breast feeding patients;
7. Allergic to a drug ingredient or component;
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival(OS) | The maximum time in follow up was approximately 12 months
  OS is defined as the time from randomization to death due to any cause, or censored at date last known alive.

SECONDARY OUTCOMES:
Progression Free Survival | The maximum time in follow up was 12 months
  Progression-free survival was defined as the time from the date of randomization to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurs first.
Objective Response Rate | Assessment every 6 weeks after initial response; maximum time on study 12 months
  Objective response rate was based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Time to Treatment Failure | The maximum time in follow up was 12 months
  Time from randomization to discontinuation of treatment for any reason, including disease progression, treatment toxicity or death.
Percentage of Patients With Tumor Marker (CA 19-9) Response | Baseline to treatment discontinuation every 6 weeks; The maximum time in follow up was 12 months
  Response was defined as a decrease of 50% of CA19-9 in relation to the baseline level at least once during the treatment period.
Quality of life（QoL） | Baseline to treatment discontinuation every 6 weeks; The maximum time in follow up was 12 months
  QoL was based on EORTC-QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Qinhuai Medical Area, General Hospital of PLA Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui J, Qin S, Zhou Y, Zhang S, Sun X, Zhang M, Cui J, Fang W, Gu K, Li Z, Wang J, Chen X, Yao J, Zhou J, Wang G, Bai Y, Xiao J, Qiu W, Wang B, Xia T, Wang C, Kong L, Yin J, Zhang T, Shen X, Fu D, Gao C, Wang H, Wang Q, Wang L. Irinotecan hydrochloride liposome HR070803 in combination with 5-fluorouracil and leucovorin in locally advanced or metastatic pancreatic ductal adenocarcinoma following prior gemcitabine-based therapy (PAN-HEROIC-1): a phase 3 trial. Signal Transduct Target Ther. 2024 Sep 19;9(1):248. doi: 10.1038/s41392-024-01948-4. PMID 39300077